CLINICAL TRIAL: NCT00580710
Title: Investigation Into the Effects Upon Brain Response to Change in Circulating Glucose Levels in Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0108012609; 2R01DK020495-37 (NIH)
Record Dates: First submitted 2007-12-19; First posted 2007-12-27 (Estimated); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Type 1 Diabetes; Hypoglycemia
Keywords: type 1 diabetes; hypoglycemia; magnetic resonance imaging
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (7):
- conventionally treated: conventionally treated, relatively poorly controlled patients with type 1 diabetes
- intensively treated: intensively treated, well controlled patients with type 1 diabetes
- lean healthy: age- and sex- matched non-diabetic, normal weight (BMI > or = 18.5 but < or = 25 kg/m2) control subjects
- obese subjects: obese individuals defined as BMI > or = 30kg/m2
- type 2 diabetics: Type 2 diabetics on diet only or diet and Metformin
- type 1 diabetes unaware: Type 1 diabetics unaware of hypoglycemic symptoms
- type 1 diabetes aware: Type 1 diabetics aware of hypoglycemic symptoms

SUMMARY:
This study is designed to investigate the effects of diabetes mellitus and its treatment upon the body's responses to low blood glucose (blood sugar) levels. Diabetes is a medical condition in which blood glucose can rise very high. Treatment of diabetes mellitus involves giving insulin (a hormone), which can occasionally cause blood glucose to fall too low. The body responds to low glucose levels by producing a number of hormones, which act against the insulin to help correct the low blood glucose. These hormones also provide symptoms which warn that the glucose is falling too far. These protective warnings by the body may be different in people with diabetes. We want to test whether this also means that diabetes changes the sensitivity of brain function to a lowering of blood glucose levels. In order to answer this question, we need to compare the response of people with diabetes with the response of people who do not have diabetes.

The plan of the study is to lower the subject's blood glucose using insulin, while measuring what changes occur in brain function using what is called functional magnetic resonance imaging (fMRI).

DETAILED DESCRIPTION:
Previous studies have shown that a person with type 1 diabetes is less likely to suffer the long term microvascular complications of diabetes (eye, kidney and nerve damage) if they strive to achieve as near normal a blood glucose as possible. Unfortunately the tighter the blood glucose control is, the more likely the subject is to suffer episodes of hypoglycemia. Hypoglycemia is often the aspect of diabetes management most feared by people with diabetes and may cause more anxiety than the threat of advanced complications.

For many people with diabetes the problem of hypoglycemia is compounded by the development of the syndrome of hypoglycemia unawareness. One aspect of hypoglycemia unawareness is impairment of the hormones normally released as blood glucose falls. Hypoglycemia triggers a release of such insulin antagonists as epinephrine, norepinephrine, glucagon, growth hormone and cortisol. These hormones act synergistically with the autonomic nervous system to raise blood glucose, counteracting insulin and restoring normoglycemia. These homeostatic mechanisms are also responsible for some of the early symptoms of low blood glucose, providing a warning to insulin-treated diabetics as glucose falls. A number of studies including research from this unit have established that strict metabolic control is associated with impairment of the normal counterregulatory response to hypoglycemia and a loss of hypoglycemia awareness.

The brain is central to the recognition of hypoglycemia and the coordination of the counterregulatory response. Neural tissue depends mainly on glucose for its energy supply. As circulating glucose falls beneath the level needed to maintain glucose transport across the blood-brain barrier, a variety of defense mechanisms are activated, including symptoms of cognitive dysfunction. However, the precise nature and causes of the adverse CNS effects of hypoglycemia are not well understood.

Functional magnetic resonance imaging (fMRI) provides a tool to measure the effects of hypoglycemia on the patterns and magnitudes of neuronal activation in the human brain, in both normal and diabetic subjects.

ELIGIBILITY:
Inclusion Criteria:

* All subjects:
* on a weight maintaining diet
* ability to read and speak English fluently
* For All Type 1 Diabetics all of the above inclusion criteria AND C-peptide negative AND no evidence of neuropathy or proliferative retinopathy
* Only for Type 1 Diabetics in the intensively treated group: HbA1c < 7.5% AND documented hypoglycemia at least once per week over at least 4 weeks of frequent daily self monitoring
* Only for Type 1 Diabetics in the conventionally treated group:HbA1c ≥ 8.5%
* Age 18-40 years in the groups 1,2, and 3. Age 18-50 in groups arm 2 obese and control.
* BMI <30 in the groups 1,2, and 3; BMI >18.4 but < or = 25 in the arm control group; and BMI > or = 30kg/m2 in the obese group.

Exclusion Criteria:

* Pregnancy
* History of neurologic or cardiovascular disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The recruited subjects will reflect the gender and ethnic distribution of the Yale and New Haven community. The recruited subjects with type 1 diabetes will reflect the demographics of the clinic population in New Haven. Subject selection is independent of race and sex.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2001-08; Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Brain response to blood glucose levels | 4 to 8 weeks
  Brain response is operationally defined as: fMRI BOLD signal to detect differences in brain activation in response to changes in glucose levels taken between 4 to 8 weeks after subject enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sherwin, M.D., Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Parikh L, Seo D, Lacadie C, Belfort-Deaguiar R, Groskreutz D, Hamza M, Dai F, Scheinost D, Sinha R, Todd Constable R, Sherwin R, Hwang JJ. Differential Resting State Connectivity Responses to Glycemic State in Type 1 Diabetes. J Clin Endocrinol Metab. 2020 Jan 1;105(1):1-13. doi: 10.1210/clinem/dgz004. PMID 31511876